CLINICAL TRIAL: NCT04069702
Title: Pilot Testing a Virtual Reality Protocol for Improving Pain and Pain-Related Distress in Patients With Advanced Stage Colorectal Cancer
Brief Title: Virtual Reality for Improving Pain and Distress in Patients With Advanced Stage Colorectal Cancer
Acronym: VR Blue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Colorado, Denver (Other); Palliative Care Research Cooperative Group (Network); National Institute of Nursing Research (NINR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103248; U2CNR014637 (NIH)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2022-08-22 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR Blue (Experimental): VR Blue is a protocol for patients with advanced stage colorectal cancer who experience persistent pain. Participants will complete a single 30-minute laboratory-based virtual reality underwater/sea environment (VR Blue) session. VR Blue is an immersive computer-generated environment featuring calming scenic graphics and relaxing nature music.
  Interventions: Behavioral: VR Blue

INTERVENTIONS:
Behavioral: VR Blue — VR Blue provides patients with an immersive computer-generated environment that can reduce pain, tension and distress.

SUMMARY:
Patients with advanced colorectal cancer often experience high levels of debilitating pain and pain-related psychological distress. Pain in cancer patients is typically treated with analgesics. There is growing agreement that non-pharmacological pain management strategies are needed to treat pain in advanced cancer patients. Recent evidence suggests Virtual Reality (VR) experiences can lead to reductions in acute pain; however, VR has not been tested in advanced cancer patients having persistent pain. VR could represent a valuable addition to our current armamentarium of treatments for persistent pain in palliative care patients. VR provides individuals with an immersive computer-generated environment that can reduce pain, tension and distress.

The proposed study builds upon and extends preliminary research in healthy participants conducted by Luana Colloca, MD, PhD. Dr. Colloca is a consultant on this project and the proposed study would be the first to extend VR Blue to a clinical population and test its effects on clinical pain. The objective is to gather initial data on advanced colorectal cancer patients' immediate response to a single VR session. The investigators will examine feasibility, acceptability, safety, and impact of exposure to VR Blue on the clinical pain experience of advanced colorectal cancer patients. The study will collect data on pain, tension and distress pre-, midpoint, and post-VR. The investigators will also examine how pre- to post-VR changes in key cognitive variables (i.e., pain catastrophizing, pain self-efficacy) relate to VR-related changes in pain, tension and distress.

The investigators will also collect qualitative data following participants' VR experience to better understand patients' preferences, thoughts and feelings about the VR experience. Data will be used to optimize VR Blue for future study, including developing an intervention to support a multi-session VR protocol for advanced colorectal cancer patients. The proposed study represents the first step in a program of clinical research that seeks to test the efficacy of VR in improving pain and pain-related symptoms in advanced colorectal cancer patients. In the proposed study, the investigators will collect quantitative and qualitative data on the impact of VR Blue on pain and pain-related outcomes in 20 advanced colorectal cancer patients.

DETAILED DESCRIPTION:
Patients with advanced colorectal cancer often experience high levels of debilitating pain and pain-related psychological distress. Pain in cancer patients is typically treated with analgesics. Unfortunately, analgesics are not uniformly effective and often are associated with poorly tolerated side effects (e.g., constipation, nausea, sedation). There is growing agreement that non-pharmacological pain management strategies are needed to treat pain in advanced cancer patients. Recent evidence suggests Virtual Reality (VR) experiences can lead to reductions in acute pain; however, VR has not been tested in advanced cancer patients having persistent pain. VR could represent a valuable addition to our current armamentarium of treatments for persistent pain in palliative care patients.

VR provides individuals with an immersive computer-generated environment that can reduce pain, tension and distress. VR may be particularly likely to positively impact cognitive pathways by changing pain-related cognitions (e.g., decreasing pain catastrophizing, increasing self-efficacy for pain control). VR-based interventions have the potential to alter these negative ways of thinking, and advanced cancer patients with persistent pain and pain-related distress may be particularly likely to benefit.

The proposed study builds upon and extends preliminary research in healthy participants conducted by Luana Colloca, MD, PhD. That study found that exposure to a 30-minute virtual underwater/sea environment (VR Blue) produced significant increases in pain tolerance for thermal pain stimuli compared to control conditions. Dr. Colloca is a consultant on this project and the proposed study would be the first to extend VR Blue to a clinical population and test its effects on clinical pain. The objective is to gather initial data on advanced colorectal cancer patients' immediate response to a single VR session. The investigators will examine feasibility, acceptability, safety, and impact of exposure to VR Blue on the clinical pain experience of advanced colorectal cancer patients. The study will collect data on pain, tension and distress pre-, midpoint, and post-VR. The investigators will also examine how pre- to post-VR changes in key cognitive variables (i.e., pain catastrophizing, pain self-efficacy) relate to VR-related changes in pain, tension and distress.

The investigators will also collect qualitative data following participants' VR experience to better understand patients' preferences, thoughts and feelings about the VR experience. Data will be used to optimize VR Blue for future study, including developing an intervention to support a multi-session VR protocol for advanced colorectal cancer patients. The proposed study represents the first step in a program of clinical research that seeks to test the efficacy of VR in improving pain and pain-related symptoms in advanced colorectal cancer patients. In the proposed study, the investigators will collect quantitative and qualitative data on the impact of VR Blue on pain and pain-related outcomes in 20 advanced colorectal cancer patients.

The long-term goal of this research is to improve quality of life in advanced colorectal cancer patients by decreasing pain, tension and distress. This project will provide preliminary data that will be used to inform and optimize development of a multi-session VR protocol to be tested in patients with advanced stage colorectal cancer that could be generalizable to other palliative care populations with pain.

ELIGIBILITY:
Inclusion Criteria:

* age 18-85
* a diagnosis of stage IV colorectal cancer
* clinical pain documented in medical chart (>4 on a 0-10 scale) and confirmed on the day of their study appointment (>4 on a 0-10 scale)
* being able to read and speak English
* self-reported normal or corrected to normal vision
* self-reported normal hearing

Exclusion Criteria:

* a serious mental illness (e.g., schizophrenia, bipolar disorder) as indicated by medical records
* a medical condition that contraindicates safe participation in the study (e.g., recent myocardial infarction)
* visual, hearing, or cognitive impairment that will interfere with the patient's ability to engage in the intervention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Kelleher, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of the NIH data sharing directive, de-identified data from this study will be transferred to the PCRC De-Identified Data Repository located at the University of Colorado. The PCRC fully supports the Final NIH Statement on Sharing Research Data, and will assist all investigators and study personnel to ensure their compliance. Consistent with OMB Circular A-110 and subsequent NIH Grants Policy Statements, the PCRC will provide access to all de-identified data collected as part of PCRC-supported investigations, insofar as access is consistent with IRB/CHR rules, local, state, and Federal laws and regulations, and the HIPAA Privacy Rule.
Supporting Information: Study Protocol
Time Frame: Data will become available after completion of the study and when summary data are published and otherwise made available. From this timepoint, data will be available for 5 years.
Access Criteria: The Principal Investigator will work with requesters and IRBs on a case by case basis.

REFERENCES:
- See also: Pre-print: Daily Lactobacillus Probiotic versus Placebo in COVID-19-Exposed Household Contacts (PROTECT-EHC): A Randomized Clinical Trial — https://www.medrxiv.org/content/10.1101/2022.01.04.21268275v1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VR Blue
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VR Blue
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Pain Right Now [Mean (Standard Deviation); unit: units on a scale] — Pain will be assessed with the Brief Pain Inventory (BPI). Patients will rate their "pain right now" from 0=no pain to 10=worst pain imaginable. An average of the responses to these items is used to create a single pain severity score.
  units on a scale | 2.8 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility, Assessed by Examining Number of Participants Accrued
Description: Feasibility was assessed by examining number of participants accrued.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | VR Blue
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: Feasibility, Assessed by Examining Number of Participants With >80% Adherence to the Protocol
Description: Feasibility will be assessed by examining protocol adherence (>80% adherence to the protocol [defined in this study as the degree to which participants are willing and able to complete the 30-minute VR exposure])
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | VR Blue
Number analyzed (Participants) | 20
Participants | 20

3. Primary Outcome: Feasibility, Assessed by Number of Participants With Completed Data
Description: Feasibility will be assessed by examining completed data (>80% data collected at the study appointment, including pre-, midpoint, and post-VR assessments)
Time Frame: 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | VR Blue
Number analyzed (Participants) | 20
Participants | 20

4. Primary Outcome: Acceptability Using the Client Satisfaction Questionnaire
Description: This questionnaire contains 10 items rated from 1=low acceptability to 4=high acceptability; scores are created by utilizing the Likert Scale to average Client Satisfaction Questionnaire answers resulting in a score range from 1-4. The participant will complete this acceptability questionnaire as part of their post-VR session assessment.
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Blue
Number analyzed (Participants) | 20
score on a scale | 3.30 (0.41)

5. Primary Outcome: Number of Participants With VR Side Effects
Description: Safety of the VR protocol will be assessed based on participants' report of VR side effects, such as motion sickness, dizziness, headache, nausea, or other negative physical reactions
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | VR Blue
Number analyzed (Participants) | 20
Participants | 20

6. Secondary Outcome: Change in Pain Severity as Assessed With the Brief Pain Inventory (BPI)
Description: Pain will be assessed with the Brief Pain Inventory (BPI). Patients will rate their "pain right now" from 0=no pain to 10=worst pain imaginable. An average of the responses to these items is used to create a single pain severity score.
Time Frame: Pre-, post-VR session, approximately 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Blue
Number analyzed (Participants) | 20
score on a scale | 1.15 (1.14)

7. Secondary Outcome: Pain Interference as Assessed With the Brief Pain Inventory (BPI) - Pain Interference Scale
Description: Pain interference will be assessed with the Brief Pain Inventory (BPI) - Pain Interference Scale. Patients will rate how much pain interfered with a variety of activities and mood states over the last 7 days from 0=does not interfere to 10=completely interferes. An average of the responses to these items is used to create a single pain severity score.
Time Frame: Pre-VR session assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Blue
Number analyzed (Participants) | 20
score on a scale | 2.86 (2.07)

8. Secondary Outcome: Change in Tension as Measured With the Visual Analog Scale (VAS)
Description: Visual Analog Scale (VAS) items are rated on a 0-100 scale. 0=no tension at all, 100=maximum tolerable tension. An average of the responses at each time-point were used to create a single score of change from pre-VR session to post-VR session.
Time Frame: Pre-, post-VR session. Full study visit starting at pre-VR and ending at Post-VR is approximately 90 minutes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Blue
Number analyzed (Participants) | 20
score on a scale | 7.70 (12.70)

9. Secondary Outcome: Change in Distress as Measured With the Visual Analog Scale (VAS)
Description: Visual Analog Scale (VAS) items are rated on a 0-100 scale. 0=no stress at all, 100=maximum tolerable stress. An average of the responses at each time-point were used to create a single score of change from pre-VR session to post-VR session.
Time Frame: Pre- and post-VR session, Full study visit starting at pre-VR and ending at Post-VR is approximately 90 minutes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Blue
Number analyzed (Participants) | 20
score on a scale | 7.60 (13.59)

10. Secondary Outcome: Change in Pain Catastrophizing as Measured With the Coping Strategies Questionnaire's Pain Catastrophizing Subscale
Description: Items will be rated on a scale ranging from 0=never do to 6=always do when in pain. An average of the responses to these items is used to create a single score of change from pre-VR session to post-VR session.
Time Frame: Pre- and post-VR session, approximately 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Blue
Number analyzed (Participants) | 20
score on a scale | 0.88 (0.89)

11. Secondary Outcome: Change in Pain Self-efficacy as Measured Using Items Adapted From the Self-efficacy for Pain Management Subscale of the Chronic Pain Self-Efficacy Scale
Description: Self-efficacy will be measured using items adapted from the self-efficacy for pain management subscale of the Chronic Pain Self-Efficacy Scale. Items are rated on a 10-point scale ranging from 10=very uncertain to 100=very certain. Scores are averaged to give an overall value of change from pre-VR session to post-VR session for pain self-efficacy.
Time Frame: Pre- and post-VR session, approximately 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VR Blue
Number analyzed (Participants) | 20
score on a scale | 72.60 (16.49)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the one-time study visit which lasted approximately 90 minutes.
Arm/Group | VR Blue
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04069702/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04069702/ICF_000.pdf